CLINICAL TRIAL: NCT05554419
Title: Eradicating Measurable Residual Disease in Patients With Acute Myeloid Leukemia (AML) Prior to StEm Cell Transplantation (ERASE): A MyeloMATCH Treatment Trial
Brief Title: Testing the Use of Combination Therapy in Patients With Persistent Low Level Acute Myeloid Leukemia Following Initial Treatment, The ERASE Study (A MyeloMATCH Treatment Trial)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-07799; NCI-2022-07799 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MM2YA-EA01 (Other: ECOG-ACRIN Cancer Research Group); MM2YA-EA01 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2022-09-23; First posted 2022-09-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Acute Myeloid Leukemia Arising From Previous Myeloproliferative Neoplasm; Acute Myeloid Leukemia Post Cytotoxic Therapy; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; Biopsy; Cytarabine; CPX-351; Daunorubicin; Injections; Liposomes; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- ARM A (cytarabine) (Active Comparator): Patients receive cytarabine IV on study. Patients undergo bone marrow aspiration and biopsy on study. Patients may also undergo ECHO and/or MUGA as clinically indicated.
  Interventions: Procedure: Bone Marrow Aspiration and Biopsy; Drug: Cytarabine; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan
- ARM B (cytarabine, venetoclax) (Experimental): Patients receive cytarabine IV and venetoclax PO on study. Patients undergo bone marrow aspiration and biopsy on study. Patients may also undergo ECHO and/or MUGA as clinically indicated.
  Interventions: Procedure: Bone Marrow Aspiration and Biopsy; Drug: Cytarabine; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Drug: Venetoclax
- ARM C (liposomal daunorubicin-cytarabine, venetoclax) (Experimental): Patients receive liposome-encapsulated daunorubicin-cytarabine IV and venetoclax PO on study. Patients undergo bone marrow aspiration and biopsy on study. Patients may also undergo ECHO and/or MUGA as clinically indicated.
  Interventions: Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Echocardiography Test; Drug: Liposome-encapsulated Daunorubicin-Cytarabine; Procedure: Multigated Acquisition Scan; Drug: Venetoclax
- ARM D (azacitidine, venetoclax) (Experimental): Patients receive azacitidine IV or SC and venetoclax PO on study. Patients undergo bone marrow aspiration and biopsy on study. Patients may also undergo ECHO and/or MUGA as clinically indicated.
  Interventions: Drug: Azacitidine; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacitidine; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
  Arms: ARM D (azacitidine, venetoclax)
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspiration and biopsy
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
  Arms: ARM A (cytarabine); ARM B (cytarabine, venetoclax)
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Liposome-encapsulated Daunorubicin-Cytarabine — Given IV
  Other Names: CPX 351; CPX-351; CPX351; Cytarabine and Daunorubicin Liposomal; Cytarabine-Daunorubicin Liposome for Injection; Daunorubicin and Cytarabine (Liposomal); Liposomal AraC-Daunorubicin CPX-351; Liposomal Cytarabine-Daunorubicin; Liposome-encapsulated Combination of Daunorubicin and Cytarabine; Vyxeos
  Arms: ARM C (liposomal daunorubicin-cytarabine, venetoclax)
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto
  Arms: ARM B (cytarabine, venetoclax); ARM C (liposomal daunorubicin-cytarabine, venetoclax); ARM D (azacitidine, venetoclax)

SUMMARY:
This phase II MyeloMATCH treatment trial compares cytarabine versus (vs.) cytarabine and venetoclax vs. liposome-encapsulated daunorubicin-cytarabine and venetoclax vs. azacitidine and venetoclax for treating patients who have residual disease after treatment for acute myeloid leukemia (AML). Cytarabine is in a class of medications called antimetabolites. It works by slowing or stopping the growth of cancer cells in the body. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Liposome-encapsulated daunorubicin-cytarabine is a drug formulation that delivers daunorubicin and cytarabine in small spheres called liposomes, which may make the drugs safer or more effective. Azacitidine is a drug that interacts with DNA and leads to the activation of tumor suppressor genes, which are genes that help control cell growth. This study may help the study doctors find out if the different drug combinations are equally effective to the usual approach of cytarabine alone while requiring a shorter duration of treatment. To decide if they are better, the study doctors will be looking to see if the study drugs lead to a higher percentage of patients achieving a deeper remission compared to cytarabine alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To improve the rate of measurable residual disease (MRD) negative complete remission (CR) in patients with acute myeloid leukemia (AML) who have achieved a MRD positive CR after induction chemotherapy received in a myeloMATCH young adult basket tier-1 protocol.

II. To determine the rate of achieving MRD negative CR after 2 cycles of post-remission therapy with cytarabine vs. cytarabine + venetoclax or liposome-encapsulated daunorubicin-cytarabine (daunorubicin and cytarabine liposome) + venetoclax azacitidine + venetoclax in AML or myelodysplastic syndrome (MDS) who were MRD positive post induction therapy.

SECONDARY OBJECTIVES:

I. To determine the disease-free survival, overall survival in this group of patients.

II. Assess the percentage of patients who receive allogeneic hematopoietic stem cell transplantation (HCT).

III. Compare toxicities of each experimental arm with the control arm.

EXPLORATORY OBJECTIVES:

I. Evaluate MRD kinetics by following patients with detectable MRD through tier 2 and beyond.

II. Evaluate longer term outcomes by treatment arm, genomics, MRD outcome, and other features as patients receive additional myeloMATCH therapies to generate testable hypotheses for more precise patient selection for these therapies aimed at improving outcomes.

OUTLINE: Patients are randomized to 1 of 4 arms.

ARM A: Patients receive cytarabine intravenously (IV) on study. Patients undergo bone marrow aspiration and biopsy on study. Patients may also undergo echocardiogram (ECHO) and/or multigated acquisition scan (MUGA) as clinically indicated.

ARM B: Patients receive cytarabine IV and venetoclax orally (PO) on study. Patients undergo bone marrow aspiration and biopsy on study. Patients may also undergo ECHO and/or MUGA as clinically indicated.

ARM C: Patients receive liposome-encapsulated daunorubicin-cytarabine IV and venetoclax PO on study. Patients undergo bone marrow aspiration and biopsy on study. Patients may also undergo ECHO and/or MUGA as clinically indicated.

ARM D: Patients receive azacitidine IV or subcutaneously (SC) and venetoclax PO on study. Patients undergo bone marrow aspiration and biopsy on study. Patients may also undergo ECHO and/or MUGA as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be >= 18 and =< 59 years of age
* Patient must have Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patient must have morphologically documented AML or secondary AML (from prior conditions such as myelodysplastic syndrome [MDS], myeloproliferative neoplasm [MPN]) or therapy related AML (t-AML), as defined by World Health Organization (WHO) criteria
* Patient must have completed induction chemotherapy in a myeloMATCH young adult tier-1 protocol. Patient may have received prior hypomethylating agents (HMAs). Patient may have received prior azacitidine + venetoclax
* Patient must have been assigned to this protocol by myeloMATCH master screening and reassessment protocol (MSRP)/MATCHBOX. Patients thereby assigned will have attained complete remission (CR) or CR with partial hematologic recovery (CRh) (defined as CR with [absolute neutrophil count (ANC)] >= 500/mcL and/or platelets > 50/mcL) with detectable MRD at time of assignment. MRD is defined as > 0.1% flow cytometry on bone marrow (BM) biopsy as assessed by MDNet. The definition of CR or CRh may be made +/- 2 weeks from BM biopsy
* Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible
* Patient must have recovered (i.e.: resolved to < grade 2) from adverse events related to prior anti-cancer therapy at the time of randomization with the exception of alopecia
* Absolute neutrophil count (ANC) >= 500/mcL (obtained =< 7 days prior to protocol randomization)
* Platelets >= 50,000/mcL (obtained =< 7 days prior to protocol randomization)
* Total bilirubin =< 2 x institutional upper limit of normal (ULN) (obtained =< 7 days prior to protocol randomization)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x institutional ULN (obtained =< 7 days prior to protocol randomization)
* Creatinine =< 1.5 x institutional ULN OR >= 50 mL/min.1.73 m^2 (obtained =< 7 days prior to protocol randomization)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of randomization are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Patients must be able to swallow oral tablets and be free of gastrointestinal (GI) absorption issues

Exclusion Criteria:

* Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used.

  * All patients of childbearing potential must have a blood test or urine study within 14 days prior to randomization to rule out pregnancy.
  * A patient of childbearing potential is defined as anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patients of childbearing potential and/or sexually active patients must not expect to conceive or father children by using an accepted and effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the study and continue for 6 months after the last dose of daunorubicin + cytarabine liposome, 6 months after the last dose of azacitidine for patients of childbearing potential, 3 months after the last dose of azacitidine for male patients, and for 30 days after the last dose of venetoclax. Patient must also abstain from nursing an infant for 2 weeks after the last dose of daunorubicin + cytarabine liposome and for 1 week after the last dose of azacitidine
* Patients must not have FLT3 TKD or ITD mutation. Patients with this mutation, will be excluded from this study because myeloMATCH plans separate studies in tier-2 for those patients
* Patient must not be receiving any other investigational agents at the time of randomization
* Patient must not have history of allergic reactions attributed to compounds of similar chemical or biologic composition to cytarabine, azacitidine, venetoclax or daunorubicin and cytarabine liposome
* Patients must not have uncontrolled intercurrent illness including but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or serious chronic gastrointestinal conditions associated with diarrhea

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 184 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of measurable residual disease (MRD) negative complete remission (CR) | Following 2 cycles of consolidation (56 days)
  Will be centrally evaluated. The MRD negative CR frequency will be compared between each experimental arm and the standard therapy arm using Fisher's exact test with one-sided alpha of 0.10 for each comparison. Test results with one-sided p-value < 0.10 will be considered statistically significant. Multivariable logistic regression modeling will also be used to examine the treatment effect between each experimental arm and the standard therapy arm, adjusting for stratification factors and other possible clinical and biological risk factors.

SECONDARY OUTCOMES:
Overall survival | Between randomization and death from any cause, assessed up to 10 years
  Estimates, including medians and confidence intervals, will be calculated using the Kaplan-Meier method. Comparison between each experimental arm and the standard therapy arm will be conducted using the one-sided log-rank test. Only nominal p-values will be provided. Cox proportional hazards models will also be used to assess the treatment effect, adjusting for stratification factors and other possible clinical and biological risk factors.
Disease-free survival | From randomization to relapse or death in remission, assessed up to 10 years
  Estimates, including medians and confidence intervals, will be calculated using the Kaplan-Meier method. Comparison between each experimental arm and the standard therapy arm will be conducted using the one-sided log-rank test. Only nominal p-values will be provided. Cox proportional hazards models will also be used to assess the treatment effect, adjusting for stratification factors and other possible clinical and biological risk factors.
Rate of allogeneic transplant | Up to 10 years
Incidence of adverse events | Up to 10 years
  Toxicity will be determined using the Common Terminology Criteria for Adverse Events (CTCAE).

CONTACTS AND LOCATIONS:
Overall Officials: Ehab L Atallah, Principal Investigator — ECOG-ACRIN Cancer Research Group

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm